CLINICAL TRIAL: NCT01225640
Title: A Phase 2a, Open-Label, Randomized Study In Treatment-Naive, Sputum Smear Positive Subjects With Drug-Sensitive Pulmonary Tuberculosis To Assess Early Bactericidal Activity (EBA) And Whole Blood Activity (WBA) Of PNU-100480 (PF-02341272)
Brief Title: PNU-100480 In Newly Diagnosed, Drug Sensitive Patients With Pulmonary TB; Early Bactericidal Activity; Whole Blood Assay
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sequella, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1171003
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; EBA; WBA
MeSH Terms: conditions — Tuberculosis | interventions — PNU-100480

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PNU-100480 600 mg BID (Experimental)
  Interventions: Drug: PNU-100480
- PNU-100480 1200 mg QD (Experimental)
  Interventions: Drug: PNU-100480
- RHZE (Active Comparator): conjugated tablet with 4 drug combination of RHZE, Rifafour® e275 will be used in countries where can be sourced locally
  Interventions: Drug: RHZE

INTERVENTIONS:
Drug: PNU-100480 — 600 mg twice daily (BID) for 14 days
  Arms: PNU-100480 600 mg BID
Drug: PNU-100480 — 1200 mg once daily (QD) for 14 days
  Arms: PNU-100480 1200 mg QD
Drug: RHZE — Combination tablet (RHZE) dosed by weight. Dosage strength per tablet is 150 mg Rifampicin (R)/75 mg Isoniazid (H)/400 mg Pyrazinamide (Z)/275 mg Ethambutol (E)
  Other Names: Rifafour, Rimstar
  Arms: RHZE

SUMMARY:
PNU-100480 is being developed for the treatment of both drug resistant and sensitive tuberculosis. This is an efficacy and safety study to characterize the effect of PNU-100480 when given for 14 days to treatment-naive patients with drug-sensitive pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females between 18 and 65 years; women of childbearing potential must be willing to adhere to lifestyle requirements regarding contraception/pregnancy prevention.
* Newly diagnosed sputum smear-positive pulmonary TB confirmed with acid-fast bacillus (AFB) smear and chest x-ray. Patients with TB more than 5 years ago who completed treatment, are healthy, and meet other inclusion criteria may be included.
* Body weight between 40 and 90 kg, inclusive (in light clothing, no shoes).
* Reasonably normal hemoglobin (>=8 gm/dL), renal function (serum creatinine <2 mg/dL), hepatic function (serum AST <3xULN and total bilirubin <1.3 mg/dL), and random glucose <150 mg/dL.

Exclusion Criteria:

* HIV infection with helper/inducer T-lymphocytes (CD4 cell) count of <=350x10-6/L.
* Presence of significant hemoptysis. Subjects who cough up frank blood (more than blood streaked sputum) will not be eligible.
* Pregnant or nursing females; females of childbearing potential unwilling or unable to adhere to contraception guidelines.
* Significant respiratory impairment (respiratory rate >35/minute).
* Clinical suspicion of disseminated TB or tuberculosis meningitis.
* Subjects with diabetes mellitus on insulin and/or who have poorly controlled disease.
* Subjects with confirmed or suspected multi-drug resistant TB.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is rate of change in sputum log CFU/mL count (EBA) from Days 0-2. | Days 0-2

SECONDARY OUTCOMES:
Rate of change in sputum log CFU/mL count (extended EBA). | Days 2-14
Rate of change in sputum log CFU/mL count (extended EBA). | Days 0-14
Rate of change in culture time to positivity (TTP) measured by MGIT and in log transformed TTP | Days 02-; 2-14; 0-14
Cumulative whole blood bactericidal activity (measured as log reduction in CFU) against intracellular M. tuberculosis relative to administered dose and drug PK | Day 1
Cumulative whole blood bactericidal activity (measured as log reduction in CFU) against intracellular M. tuberculosis relative to administered dose and drug PK | Day 13-14
Plasma concentrations of PNU-100480 and PNU-101603 will be used to determine PK parameters (AUCtau, AUC tau,ss, Cmax, Tmax, terminal half-life t1/2, Cavg, Rac) as data permit | Day 1
Plasma concentrations of PNU-100480 and PNU-101603 will be used to determine PK parameters (AUCtau, AUC tau,ss, Cmax, Tmax, terminal half-life t1/2, Cavg, Rac) as data permit | Day 13-14
Safety assessments including physical exams, AEs, laboratory tests, ECGs, and vital signs. | Phys exam, AEs, and vitals are done at every visit (Screening through Day 15, Day 42/Follow-up)
Safety assessments including physical exams, AEs, laboratory tests, ECGs, and vital signs. | ECGs are done at Screening, Day 1, Day 14, 15 and 42/Follow-up
Safety assessments including physical exams, AEs, laboratory tests, ECGs, and vital signs. | Lab tests at Screening, Day 1, Day 15 and 42/Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beth Ferstenberg, M.D., Study Director — Sequella, Inc.
Locations (2):
- South Africa (2):
  - Pfizer Investigational Site, Bellville, Cape Town
  - Pfizer Investigational Site, Cape Town

REFERENCES:
- [Derived] Wallis RS, Dawson R, Friedrich SO, Venter A, Paige D, Zhu T, Silvia A, Gobey J, Ellery C, Zhang Y, Eisenach K, Miller P, Diacon AH. Mycobactericidal activity of sutezolid (PNU-100480) in sputum (EBA) and blood (WBA) of patients with pulmonary tuberculosis. PLoS One. 2014 Apr 14;9(4):e94462. doi: 10.1371/journal.pone.0094462. eCollection 2014. PMID 24732289